CLINICAL TRIAL: NCT02902315
Title: Vitamins C and E Combined With Cryotherapy on the Pain, Oxidative Stress and Inflammatory Response After Resistance Exercise Session in Untrained Volunteers
Brief Title: Antioxidants Combined With Cryotherapy on Inflammatory Response After Resistance Exercise in Untrained Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Luis Ulisses Signori, PhD, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UFSantaMaria2
Record Dates: First submitted 2016-08-19; First posted 2016-09-15 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Inflammation; Oxidative Stress; Pain
Keywords: Muscle soreness; Free radicals; Ascorbic acid; Alpha-Tocopherol; Cryotherapy; Exercise tolerance; Resistance training
MeSH Terms: conditions — Inflammation; Pain; Myalgia | interventions — Cryotherapy; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1ª Session of resistance exercises (Active Comparator): Exercise session are based on previous studies (TEIXEIRA et al., 2012; TEIXEIRA et al., 2014) and will be randomized according to the sequence of exercises (extensor bench, squat and leg press) and the interventions by drawing sealed brown envelopes. Forty minutes before basal blood collection and of the exercise session the volunteers will receive placebo (two pills wheat flour) and the remaining procedures will be conserved. The exercise sessions were comprised of four series of 10 maximum repetitions, with an interval of one minute between series and two minutes between exercises. Before the 10 maximum repetitions test and data collection, standard instructions will be given concerning the experimental procedure and execution technique of the exercises.
  Interventions: Other: Cryotherapy; Other: Vitamins C and E; Other: Vitamins C and E associated with cryotherapy; Other: Placebo
- 2ª Session of resistance exercises (Active Comparator): Exercise session are based on previous studies (TEIXEIRA et al., 2012; TEIXEIRA et al., 2014) and will be randomized according to the sequence of exercises (extensor bench, squat and leg press) and the interventions by drawing sealed brown envelopes. Forty minutes before basal blood collection and of the exercise session the volunteers will receive placebo (two pills wheat flour) and the remaining procedures will be conserved. The exercise sessions were comprised of four series of 10 maximum repetitions, with an interval of one minute between series and two minutes between exercises. Before the 10 maximum repetitions test and data collection, standard instructions will be given concerning the experimental procedure and execution technique of the exercises.
  Interventions: Other: Cryotherapy; Other: Vitamins C and E; Other: Vitamins C and E associated with cryotherapy; Other: Placebo
- 3ª Session of resistance exercises (Active Comparator): Exercise session are based on previous studies (TEIXEIRA et al., 2012; TEIXEIRA et al., 2014) and will be randomized according to the sequence of exercises (extensor bench, squat and leg press) and the interventions by drawing sealed brown envelopes. Forty minutes before basal blood collection and of the exercise session the volunteers will receive placebo (two pills wheat flour) and the remaining procedures will be conserved. The exercise sessions were comprised of four series of 10 maximum repetitions, with an interval of one minute between series and two minutes between exercises. Before the 10 maximum repetitions test and data collection, standard instructions will be given concerning the experimental procedure and execution technique of the exercises.
  Interventions: Other: Cryotherapy; Other: Vitamins C and E; Other: Vitamins C and E associated with cryotherapy; Other: Placebo
- 4ª Session of resistance exercises (Active Comparator): Exercise session are based on previous studies (TEIXEIRA et al., 2012; TEIXEIRA et al., 2014) and will be randomized according to the sequence of exercises (extensor bench, squat and leg press) and the interventions by drawing sealed brown envelopes. Forty minutes before basal blood collection and of the exercise session the volunteers will receive placebo (two pills wheat flour) and the remaining procedures will be conserved. The exercise sessions were comprised of four series of 10 maximum repetitions, with an interval of one minute between series and two minutes between exercises. Before the 10 maximum repetitions test and data collection, standard instructions will be given concerning the experimental procedure and execution technique of the exercises.
  Interventions: Other: Cryotherapy; Other: Vitamins C and E; Other: Vitamins C and E associated with cryotherapy; Other: Placebo

INTERVENTIONS:
Other: Cryotherapy — The intervention will consist of the application of hypothermia by immersion of the lower limbs of water on individuals to 15ºC for a period of 10 minutes immediately after the exercise protocol.
  Other Names: Hypothermia
Other: Vitamins C and E — The session of resistance exercises with intervention will be based on the supplementation with vitamin C (1000 mg) and vitamin E (800 IU) by oral intake (100mL of water) 40 minutes before basal blood collection.
  Other Names: Ascorbic acid; alfa-tocopherol
Other: Vitamins C and E associated with cryotherapy — The session of resistance exercises with intervention will be based on the supplementation with vitamin C (1000 mg) and vitamin E (800 IU) by oral intake (100mL of water) 40 minutes before basal blood collection. The intervention will consist of the application of hypothermia by immersion of the lower limbs of water on individuals to 15ºC for a period of 10 minutes immediately after the exercise protocol.
  Other Names: Vitamins C and E; Hypothermia
Other: Placebo — The volunteers from placebo exercise session will receive two pills (containing wheat flour) and the remaining procedures were conserved.
  Other Names: Control

SUMMARY:
Acutely resistance exercise induces inflammatory responses and leukocytosis arising of oxidative stress, that clinically manifested by pain and/or delayed onset muscle soreness (DOMS). Beginners in resistance exercise programs are more vulnerable to the effects of oxidative stress as they exhibit lower antioxidant capacity, greater lipid peroxidation and present increased perception of pain after exercises that may lead to abandonment the exercises practice. Vitamins C and E are exogenous antioxidants which are able to prevent damages caused by oxidative stress. Cryotherapy decreases temperature and reduced generation of reactive oxygen species. The aim of the present research are to investigate the effects of the concomitant of vitamins and of cryotherapy on leukocytosis, inflammatory markers, oxidative stress parameters and pain in untrained individuals submitted to a resistance exercise session.

DETAILED DESCRIPTION:
The regular practice of physical exercises promotes anti-inflammatory effects, which reduces the mortality from all causes, especially by cardiovascular diseases. On the other hand, physical exercise induces acute inflammatory responses. Acute resistance exercises provoke mechanical and metabolic stress which may vary depending on the intensity, specificity, volume and workload. During these exercises, reactive oxygen and nitrogen species (RONS) are formed and, when its production exceeds the antioxidant enzymatic capacity (Superoxide dismutase, Catalase and Glutathione peroxidase) and non-enzymatic capacity (vitamins A, C, E and uric acid) results in oxidation of cell constituents. This state of oxidative stress promotes one inflammatory response, activation and mobilization of circulating white blood cells and induce a transitory leukocytosis, that are observed during and immediately after resistance exercises. The local neutrophilia induces the amplification of inflammatory response by feedback resulting in activation and/or mobilization of the more white blood cells. This sequence of physiological events leads to muscular remodeling although, during such process, occur functional insufficiency and the sensation of pain and/or delayed onset muscular soreness (DOMS), which deserves special attention, once may lead to interruption or abandonment of exercises, especially concerning beginners in this practice.

Numerous preventive approaches have been studied intending to minimize the inflammatory response caused by resistance exercises, including the supplementation with vitamins C (ascorbic acid) and E (alfa-tocopherol). These vitamins are exogenous antioxidants which are able to prevent damages caused by RONS and consequently attenuate the oxidative damage induced by resistance exercises. Cryotherapy is defined as the therapeutic application of any substance that removes heat from the body, thus lowering the temperature of tissues. Immersion in cold water (≤ 15ºC) is a common method of heat reduction. Cryotherapy attenuates microvascular dysfunction, and decreases temperature, metabolism and oxygen demand in the electron transport chain. As a consequence, lower amounts of RONS are produced less damage was caused to adjacent molecules. The aim of the present research are to investigate the effects of the concomitant supplementation of vitamins (C and E) and cryotherapy (immersion in water at 15ºC) on leukocytosis, inflammatory markers, oxidative stress parameters and pain in untrained individuals submitted to a resistance exercise session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 35 years, body mass index (MBI: kg/m2) lower than 30, non-smokers, did not practice physical and/or regular physical exercises (less than two times per week), presented no previous diagnosis of chronic diseases (rheumatic, cardiovascular, metabolic, neurological, oncologic, immunological or hematologic disorders), is not engaged in any diet programs and is not making use of medication.

Exclusion Criteria:

* Inflammatory response (ultrasensitive C reactive protein >3 mg/dL), hyperglycemia (>100 mg/dL), leukocytosis, hyperthermia (>38ºC), changes in the systemic blood pressure (>140/90 mmHg) and/or any symptom of pain or discomfort

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Delayed onset muscle soreness (points) | Assessed 24 hours after resistance exercise session
  Twenty-four hours after the exercise session, the pain or delayed onset muscle soreness (DOMS) was evaluated by visual analog scale (0 - 10 points).

SECONDARY OUTCOMES:
Erythrocytes (/ mm3) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Blood count (/ mm3).
Platelets (/ mm3) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Blood count (/ mm3).
Leukogram (/ mm3) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Differential white blood cell counts (/ mm3). Total leukocytes, segmented neutrophils, young neutrophils (rods), monocytes, lymphocytes and eosinophils.
C reactive protein (mg/dL) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Inflammatory markers
Creatine kinase (U/L) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Inflammatory markers
Lactate dehydrogenase (mmol/L) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Inflammatory markers
Fibrinogen (mg/dL) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Inflammatory markers.
Reactive oxygen species (ROS = relative area) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Oxidative stress parameters: damage molecular.
Anti-oxidant capacity against peroxyl radicals (ACAP = deference of the areas (wtih ABAP / without ABAP) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Oxidative stress parameters: damage molecular , anti-oxidant capacity against peroxyl radicals (ACAP = deference of the areas (wtih ABAP / without ABAP)
Superoxide dismutase (SOD = units / mg protein) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Oxidative stress parameters: enzymatic molecular defense
Catalase (units / mg protein) | Baseline (before), and at 0, 30 and 120 minutes after exercises.
  Oxidative stress parameters: enzymatic molecular defense

CONTACTS AND LOCATIONS:
Overall Officials: Luis U Signori, PhD, Principal Investigator — Universidade Federal de Santa Maria
Locations (1):
- Universidade Federal do Rio Grande, Rio Grande, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvalho N, Puntel G, Correa P, Gubert P, Amaral G, Morais J, Royes L, da Rocha J, Soares F. Protective effects of therapeutic cold and heat against the oxidative damage induced by a muscle strain injury in rats. J Sports Sci. 2010 Jul;28(9):923-35. doi: 10.1080/02640414.2010.481722. PMID 20544483
- [Background] Nadler SF, Weingand K, Kruse RJ. The physiologic basis and clinical applications of cryotherapy and thermotherapy for the pain practitioner. Pain Physician. 2004 Jul;7(3):395-9. PMID 16858479
- [Background] Bryer SC, Goldfarb AH. Effect of high dose vitamin C supplementation on muscle soreness, damage, function, and oxidative stress to eccentric exercise. Int J Sport Nutr Exerc Metab. 2006 Jun;16(3):270-80. doi: 10.1123/ijsnem.16.3.270. PMID 16948483
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Hudson MB, Hosick PA, McCaulley GO, Schrieber L, Wrieden J, McAnulty SR, Triplett NT, McBride JM, Quindry JC. The effect of resistance exercise on humoral markers of oxidative stress. Med Sci Sports Exerc. 2008 Mar;40(3):542-8. doi: 10.1249/MSS.0b013e31815daf89. PMID 18379219
- [Background] Malm C, Nyberg P, Engstrom M, Sjodin B, Lenkei R, Ekblom B, Lundberg I. Immunological changes in human skeletal muscle and blood after eccentric exercise and multiple biopsies. J Physiol. 2000 Nov 15;529 Pt 1(Pt 1):243-62. doi: 10.1111/j.1469-7793.2000.00243.x. PMID 11080266
- [Background] Finaud J, Lac G, Filaire E. Oxidative stress : relationship with exercise and training. Sports Med. 2006;36(4):327-58. doi: 10.2165/00007256-200636040-00004. PMID 16573358
- [Background] Lewis PB, Ruby D, Bush-Joseph CA. Muscle soreness and delayed-onset muscle soreness. Clin Sports Med. 2012 Apr;31(2):255-62. doi: 10.1016/j.csm.2011.09.009. Epub 2011 Nov 23. PMID 22341015
- [Background] Nakajima T, Kurano M, Hasegawa T, Takano H, Iida H, Yasuda T, Fukuda T, Madarame H, Uno K, Meguro K, Shiga T, Sagara M, Nagata T, Maemura K, Hirata Y, Yamasoba T, Nagai R. Pentraxin3 and high-sensitive C-reactive protein are independent inflammatory markers released during high-intensity exercise. Eur J Appl Physiol. 2010 Nov;110(5):905-13. doi: 10.1007/s00421-010-1572-x. Epub 2010 Jul 17. PMID 20640440
- [Background] Rietjens SJ, Beelen M, Koopman R, VAN Loon LJ, Bast A, Haenen GR. A single session of resistance exercise induces oxidative damage in untrained men. Med Sci Sports Exerc. 2007 Dec;39(12):2145-51. doi: 10.1249/mss.0b013e318157936d. PMID 18046185
- [Background] Silva LA, Pinho CA, Silveira PC, Tuon T, De Souza CT, Dal-Pizzol F, Pinho RA. Vitamin E supplementation decreases muscular and oxidative damage but not inflammatory response induced by eccentric contraction. J Physiol Sci. 2010 Jan;60(1):51-7. doi: 10.1007/s12576-009-0065-3. Epub 2009 Oct 27. PMID 19859781
- [Background] Teixeira ADO, Franco OS, Borges MM, et al.. The importance of adjustments for changes in plasma volume in the interpretation of hematological and inflmmatory responses after resistance exercise. J Exerc Physiol 17:72-83, 2014.
- [Background] Teixeira ADO, Paulitsch FDS, Umpierre MDM, et al.. Inflammatory response after session of resistance exercises in untrained volunteers. Acta Sci Heal Sci 37:31-39, 2015. doi: 10.4025/actascihealthsci.v37i1.24149
- [Background] Schaser KD, Disch AC, Stover JF, Lauffer A, Bail HJ, Mittlmeier T. Prolonged superficial local cryotherapy attenuates microcirculatory impairment, regional inflammation, and muscle necrosis after closed soft tissue injury in rats. Am J Sports Med. 2007 Jan;35(1):93-102. doi: 10.1177/0363546506294569. Epub 2006 Dec 1. PMID 17197574
- [Background] Traber MG, Stevens JF. Vitamins C and E: beneficial effects from a mechanistic perspective. Free Radic Biol Med. 2011 Sep 1;51(5):1000-13. doi: 10.1016/j.freeradbiomed.2011.05.017. Epub 2011 May 25. PMID 21664268
- [Background] Wilcock IM, Cronin JB, Hing WA. Physiological response to water immersion: a method for sport recovery? Sports Med. 2006;36(9):747-65. doi: 10.2165/00007256-200636090-00003. PMID 16937951